CLINICAL TRIAL: NCT04530630
Title: The Efficacy, Safety, and Tolerability of Switching to a Bictegravir (BIC)/Emtricitabine(FTC)/Tenofovir Alafenamide (TAF) Regimen in Virally Suppressed Human Immunodeficiency Viruses (HIV)-Positive Patients Post-Renal Transplant
Brief Title: Switch to Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF) After Renal Transplant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-01021384
Record Dates: First submitted 2020-08-24; First posted 2020-08-28 (Actual); Results first posted 2025-08-12 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-07

CONDITIONS: HIV Infections; Renal Transplant Rejection
Keywords: HIV Positive; Post Renal Transplant; Bictegravir/Emtricitabine/Tenofovir Alafenamide; Antiretroviral; Biktarvy
MeSH Terms: conditions — HIV Infections; HIV Seropositivity | interventions — bictegravir, emtricitabine, tenofovir alafenamide, drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF) (Experimental): Participants receive a BIC/F/TAF tablet orally once daily with or without food.
  Interventions: Drug: BIC/F/TAF 50Mg-200Mg-25Mg Tablet

INTERVENTIONS:
Drug: BIC/F/TAF 50Mg-200Mg-25Mg Tablet — A three-drug fixed dose combination tablet containing 50mg of bictegravir, 200mg of emtricitabine, and 25mg of tenofovir alafenamide.
  Other Names: Biktarvy

SUMMARY:
This is an open-label study, where participants will be switched from their current HIV medication to the study drug, BIC/F/TAF. Open-label means both the investigator and the participant will know what drug will be given. Participants will be followed for 48 weeks in order to monitor the efficacy, safety and tolerability of BIC/F/TAF. The investigator hypothesizes that BIC/F/TAF will be an important addition to the management of HIV-positive post renal transplant patients, especially since it is a one pill daily dosing regimen, thereby decreasing the pill burden in this population.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old on day of signing informed consent
* Positive for human immunodeficiency virus (HIV)
* Received a previous renal transplant
* Must have controlled HIV infection for at least 3 months prior to enrollment

Exclusion Criteria:

* Received a kidney from a donor who was HIV positive (unless a false positive)
* Currently taking BIC/F/TAF for treatment of HIV
* Has allergies to any of the HIV medications in BIC/F/TAF (bictegravir, emtricitabine, or tenofovir alafenamide)
* Currently taking dofetilide or rifampin
* Is pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-11-09 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Catherine B Small, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Molina JM, Ward D, Brar I, Mills A, Stellbrink HJ, Lopez-Cortes L, Ruane P, Podzamczer D, Brinson C, Custodio J, Liu H, Andreatta K, Martin H, Cheng A, Quirk E. Switching to fixed-dose bictegravir, emtricitabine, and tenofovir alafenamide from dolutegravir plus abacavir and lamivudine in virologically suppressed adults with HIV-1: 48 week results of a randomised, double-blind, multicentre, active-controlled, phase 3, non-inferiority trial. Lancet HIV. 2018 Jul;5(7):e357-e365. doi: 10.1016/S2352-3018(18)30092-4. Epub 2018 Jun 18. PMID 29925489
- [Background] Gallant J, Lazzarin A, Mills A, Orkin C, Podzamczer D, Tebas P, Girard PM, Brar I, Daar ES, Wohl D, Rockstroh J, Wei X, Custodio J, White K, Martin H, Cheng A, Quirk E. Bictegravir, emtricitabine, and tenofovir alafenamide versus dolutegravir, abacavir, and lamivudine for initial treatment of HIV-1 infection (GS-US-380-1489): a double-blind, multicentre, phase 3, randomised controlled non-inferiority trial. Lancet. 2017 Nov 4;390(10107):2063-2072. doi: 10.1016/S0140-6736(17)32299-7. Epub 2017 Aug 31. PMID 28867497
- [Background] Sax PE, DeJesus E, Crofoot G, Ward D, Benson P, Dretler R, Mills A, Brinson C, Peloquin J, Wei X, White K, Cheng A, Martin H, Quirk E. Bictegravir versus dolutegravir, each with emtricitabine and tenofovir alafenamide, for initial treatment of HIV-1 infection: a randomised, double-blind, phase 2 trial. Lancet HIV. 2017 Apr;4(4):e154-e160. doi: 10.1016/S2352-3018(17)30016-4. Epub 2017 Feb 15. PMID 28219610
- [Background] Orkin C, Molina JM, Negredo E, Arribas JR, Gathe J, Eron JJ, Van Landuyt E, Lathouwers E, Hufkens V, Petrovic R, Vanveggel S, Opsomer M; EMERALD study group. Efficacy and safety of switching from boosted protease inhibitors plus emtricitabine and tenofovir disoproxil fumarate regimens to single-tablet darunavir, cobicistat, emtricitabine, and tenofovir alafenamide at 48 weeks in adults with virologically suppressed HIV-1 (EMERALD): a phase 3, randomised, non-inferiority trial. Lancet HIV. 2018 Jan;5(1):e23-e34. doi: 10.1016/S2352-3018(17)30179-0. Epub 2017 Oct 6. PMID 28993180
- [Background] Pozniak A, Arribas JR, Gathe J, Gupta SK, Post FA, Bloch M, Avihingsanon A, Crofoot G, Benson P, Lichtenstein K, Ramgopal M, Chetchotisakd P, Custodio JM, Abram ME, Wei X, Cheng A, McCallister S, SenGupta D, Fordyce MW; GS-US-292-0112 Study Team. Switching to Tenofovir Alafenamide, Coformulated With Elvitegravir, Cobicistat, and Emtricitabine, in HIV-Infected Patients With Renal Impairment: 48-Week Results From a Single-Arm, Multicenter, Open-Label Phase 3 Study. J Acquir Immune Defic Syndr. 2016 Apr 15;71(5):530-7. doi: 10.1097/QAI.0000000000000908. PMID 26627107
- [Background] Deeks ED. Bictegravir/Emtricitabine/Tenofovir Alafenamide: A Review in HIV-1 Infection. Drugs. 2018 Nov;78(17):1817-1828. doi: 10.1007/s40265-018-1010-7. PMID 30460547
- [Background] Eron JJ, Lelievre J-D, Kalayjian R, Slim J, et al. Safety and Efficacy of E/C/F/TAF in HIV-Infected Adults on Chronic Hemodialysis (Abstract, poster 732 presented at CROI 2018).
- [Background] Stock PG, Barin B, Murphy B, Hanto D, Diego JM, Light J, Davis C, Blumberg E, Simon D, Subramanian A, Millis JM, Lyon GM, Brayman K, Slakey D, Shapiro R, Melancon J, Jacobson JM, Stosor V, Olson JL, Stablein DM, Roland ME. Outcomes of kidney transplantation in HIV-infected recipients. N Engl J Med. 2010 Nov 18;363(21):2004-14. doi: 10.1056/NEJMoa1001197. PMID 21083386
- [Background] Locke JE, Mehta S, Reed RD, MacLennan P, Massie A, Nellore A, Durand C, Segev DL. A National Study of Outcomes among HIV-Infected Kidney Transplant Recipients. J Am Soc Nephrol. 2015 Sep;26(9):2222-9. doi: 10.1681/ASN.2014070726. Epub 2015 Mar 19. PMID 25791727
- [Background] Gunawardana M, Remedios-Chan M, Miller CS, Fanter R, Yang F, Marzinke MA, Hendrix CW, Beliveau M, Moss JA, Smith TJ, Baum MM. Pharmacokinetics of long-acting tenofovir alafenamide (GS-7340) subdermal implant for HIV prophylaxis. Antimicrob Agents Chemother. 2015 Jul;59(7):3913-9. doi: 10.1128/AAC.00656-15. Epub 2015 Apr 20. PMID 25896688
- [Background] Kraft JC, McConnachie LA, Koehn J, Kinman L, Collins C, Shen DD, Collier AC, Ho RJ. Long-acting combination anti-HIV drug suspension enhances and sustains higher drug levels in lymph node cells than in blood cells and plasma. AIDS. 2017 Mar 27;31(6):765-770. doi: 10.1097/QAD.0000000000001405. PMID 28099191
- [Background] Pharmacoeconomic Review Report: Bictegravir/Emtricitabine/Tenofovir Alafenamide (B/FTC/TAF) (Biktarvy): (Gilead Sciences Canada, Inc.): Indication: A complete regimen for the treatment of HIV-1 infection in adults with no known substitution associated with resistance the individual components of Biktarvy [Internet]. Ottawa (ON): Canadian Agency for Drugs and Technologies in Health; 2018 Oct. Available from http://www.ncbi.nlm.nih.gov/books/NBK539546/ PMID 30958667
- [Background] Castillo-Mancilla JR, Zheng JH, Rower JE, Meditz A, Gardner EM, Predhomme J, Fernandez C, Langness J, Kiser JJ, Bushman LR, Anderson PL. Tenofovir, emtricitabine, and tenofovir diphosphate in dried blood spots for determining recent and cumulative drug exposure. AIDS Res Hum Retroviruses. 2013 Feb;29(2):384-90. doi: 10.1089/AID.2012.0089. Epub 2012 Oct 10. PMID 22935078
- [Background] Castillo-Mancilla J, Seifert S, Campbell K, Coleman S, McAllister K, Zheng JH, Gardner EM, Liu A, Glidden DV, Grant R, Hosek S, Wilson CM, Bushman LR, MaWhinney S, Anderson PL. Emtricitabine-Triphosphate in Dried Blood Spots as a Marker of Recent Dosing. Antimicrob Agents Chemother. 2016 Oct 21;60(11):6692-6697. doi: 10.1128/AAC.01017-16. Print 2016 Nov. PMID 27572401
- [Background] Zheng JH, Guida LA, Rower C, Castillo-Mancilla J, Meditz A, Klein B, Kerr BJ, Langness J, Bushman L, Kiser J, Anderson PL. Quantitation of tenofovir and emtricitabine in dried blood spots (DBS) with LC-MS/MS. J Pharm Biomed Anal. 2014 Jan;88:144-51. doi: 10.1016/j.jpba.2013.08.033. Epub 2013 Aug 31. PMID 24055850
- [Background] Anderson PL, Kiser JJ, Gardner EM, Rower JE, Meditz A, Grant RM. Pharmacological considerations for tenofovir and emtricitabine to prevent HIV infection. J Antimicrob Chemother. 2011 Feb;66(2):240-50. doi: 10.1093/jac/dkq447. Epub 2010 Nov 30. PMID 21118913

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Started | 20
Completed | 19
Not Completed | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 16
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 16
  White | 1
  More than one race | 3
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Plasma HIV-1 Ribonucleic Acid (RNA) <50 Copies/ml
Description: HIV viral loads will be obtained from lab reports.
Time Frame: Up to week 48 (End of Study)
Population: One subject was excluded from data analysis due to early study withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
Participants | 19

2. Primary Outcome: Safety (Tolerability) as Measured by the Number of Subjects Who Had a Serious Adverse Event (SAE)
Time Frame: Up to week 48 (End of study)
Population: One subject was excluded from data analysis due to early withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 20
Participants | 1

3. Primary Outcome: Intracellular TAF Levels as Measured by Dried Blood Spot
Description: Fmol/punch refers to the concentration of a substance, measured in femtomoles per a specific size of a dried blood spot (DBS) punch.
Time Frame: 12 weeks
Population: One subject was excluded from data analysis due to early withdrawal.
Measure: Geometric Mean (95% Confidence Interval); unit: Femtomole (fmol)/punch of DBS
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
Femtomole (fmol)/punch of DBS
  Tenofovir-diphosphate (TFV-DP) | 1.71 [1.29 to 2.25]
  Emtricitabine triphosphate (FTC-TP) | 1.18 [0.88 to 1.59]

4. Primary Outcome: Intracellular TAF Levels as Measured by Peripheral Blood Mononuclear Cells (PBMCs)
Description: pmol/10^6 cells refers to the amount of a particular substance (in picomoles) per one million cells
Time Frame: 12 weeks
Population: One subject was excluded from data analysis due to early withdrawal.
Measure: Geometric Mean (95% Confidence Interval); unit: pmol/10^6 cells
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
pmol/10^6 cells
  TFV-DP | 2.87 [2.00 to 4.12]
  FTC-TP | 2.76 [1.85 to 4.12]

5. Primary Outcome: Renal Function as Measured by Blood Urea Nitrogen (BUN)
Time Frame: 24 weeks, 48 weeks (End of study)
Population: One subject was excluded from data analysis due to early withdrawal.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
mg/dL
  week 24 | 25.21 (9.06)
  week 48 | 23.47 (9.62)

6. Primary Outcome: Renal Function as Measured by Creatinine
Time Frame: 24 weeks, 48 weeks (End of study)
Population: One subject was excluded from data analysis due to early withdrawal.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
mg/dL
  week 24 | 1.61 (0.52)
  week 48 | 1.57 (0.52)

7. Primary Outcome: Renal Function as Measured by Creatinine Clearance
Time Frame: 24 weeks, 48 weeks (End of study)
Population: One subject was excluded from data analysis due to early withdrawal.
Measure: Mean (Standard Deviation); unit: mL/min
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
mL/min
  Week 24 | 58.10 (15.92)
  week 48 | 60.68 (15.78)

8. Primary Outcome: Renal Function as Measured by Estimated Glomerular Filtration Rate (eGFR)
Time Frame: 24 weeks, 48 weeks (End of study)
Population: One subject was excluded from data analysis due to early withdrawal.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
mL/min/1.73m^2
  week 24 | 48.32 (13.98)
  week 48 | 49.21 (14.84)

9. Primary Outcome: Tacrolimus Levels
Time Frame: 12 weeks, 24 weeks, 48 weeks (End of study)
Population: One subject was excluded from data analysis due to early withdrawal.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
ng/mL
  week 12 | 6.37 (1.78)
  week 24 | 7.97 (3.29)
  week 48 | 6.64 (2.60)

10. Secondary Outcome: Change From Baseline CD4+ T Lymphocyte Numbers Post Renal Transplant
Description: Number of CD4+ T lymphocyte counts will be obtained from lab reports
Time Frame: Day 1 (Baseline), Week 4, Week 12, Week 24, Week 36, Week 48 (End of study)
Population: 1 participant was excluded from data analysis due to early withdrawal.
Measure: Mean (Full Range); unit: cells/µL
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
cells/µL
  Baseline | 256.5263 [19 to 680]
  Week 4 | 305.8333 [24 to 1033]
  Week 12 | 342.2105 [35 to 920]
  Week 24 | 374.8947 [38 to 887]
  Week 36 | 404.6667 [103 to 958]
  Week 48 (End of Study) | 382.4211 [129 to 1174]

11. Secondary Outcome: Change From Baseline CD4+ T Lymphocyte Percentages Post Renal Transplant
Description: CD4+ T lymphocyte percentages will be obtained from lab reports
Time Frame: Day 1 (Baseline), Week 4, Week 12, Week 24, Week 36, Week 48 (End of study)
Population: 1 participant was excluded from data analysis due to early withdrawal.
Measure: Mean (Full Range); unit: Percentage of CD4+ lymphocytes
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
Percentage of CD4+ lymphocytes
  Baseline | 22.6842 [6 to 51]
  Week 4 | 25.667 [8 to 54]
  Week 12 | 25.7368 [8 to 53]
  Week 24 | 27.0526 [9 to 50]
  Week 36 | 28.1111 [10 to 56]
  Week 48 (End of Study) | 26.1579 [10 to 54]

12. Secondary Outcome: Number of Subjects With Rejection of the Kidney Transplant, Post Renal Transplant
Description: Data for kidney graft rejection will be extracted from biopsy confirmed rejections.
Time Frame: up to 48 weeks (End of study)
Population: 1 participant was excluded from data analysis due to early withdrawal.
Measure: Count of Participants; unit: Participants
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
Participants | 0

13. Secondary Outcome: Participant Satisfaction With Reduced Pill Burden and Adverse Events (Tolerability) Measured by the Health-related Quality of Life Questionnaire
Description: Satisfaction will be measured by the self-reporting health-related quality of life questionnaire ranging from 0 to 6 with higher scores indicating greater satisfaction with Biktarvy.
Time Frame: Week 24, Week 48 (End of study)
Population: One subject was excluded from data analysis due to early withdrawal.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
Number analyzed (Participants) | 19
score on a scale
  Week 24 | 5.85 [0 to 6]
  Week 48 | 5.89 [0 to 6]

ADVERSE EVENTS:
Time Frame: Up to week 48 (End of study)
Arm/Group | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF)
All-Cause Mortality (participants affected / at risk) | 0/20
Serious Adverse Events (participants affected / at risk) | 1/20
Other Adverse Events (participants affected / at risk) | 5/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF) (N=20)
Anaphylaxis (Immune system disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Bictegravir/Emtricitabine/Tenofovir Alafenamide (BIC/F/TAF) (N=20)
Loose Stool/ Diarrhea (Gastrointestinal disorders) | 5

LIMITATIONS AND CAVEATS:
The sample size was not sufficient for the statistical analysis plan as written, and, therefore, only descriptive statistics can be presented for the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-03-15): https://cdn.clinicaltrials.gov/large-docs/30/NCT04530630/Prot_SAP_000.pdf